CLINICAL TRIAL: NCT01432262
Title: A Phase 3, Open Label, Single Arm, Multicenter, Trial to Assess The Safety, Tolerability And Immunogenicity Of 13-Valent Pneumococcal Conjugate Vaccine In Healthy Adults Aged => 50 Years of Age Who Are Naive To 23-Valent Pneumococcal Polysaccharide Vaccine in Mexico.
Brief Title: 13-valent Pneumococcal Conjugate Vaccine Study in Adults => 50 Years of Age in Mexico
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B1851048; 6115A1-3020
Record Dates: First submitted 2011-06-22; First posted 2011-09-12 (Estimated); Results first posted 2013-01-08 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Pneumococcal Infections
Keywords: prevention of pneumococcal diseases
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): => 65 years of age
  Interventions: Biological: vaccine-13vPnC
- Group 2 (Experimental): 50 to 64 years of age
  Interventions: Biological: vaccine-13vPnC

INTERVENTIONS:
Biological: vaccine-13vPnC — Single dose of 0.5 ml of 13vPnC administered in deltoid muscle of arm at visit 1 (day 1)
  Other Names: 13-valent pneumococcal conjugate vaccine
  Arms: Group 1
Biological: vaccine-13vPnC — Single dose of 0.5 ml of 13vPnC administered in deltoid muscle of arm at visit 1 (day 1)
  Other Names: 13-valent pneumococcal conjugate vaccine
  Arms: Group 2

SUMMARY:
The purpose of this study will be to assess the safety, tolerability, and immunogenicity of 13-Valent Pneumococcal Conjugate Vaccine (13vPnC) when given to healthy adults older than 50 years of age who haven't received 23-valent pneumococcal polysaccharide vaccine in Mexico.

ELIGIBILITY:
Inclusion Criteria:

* Male or female older than 50 years of age
* Eligibility must be determined by medical history, physical exam and clinical judgment
* Able to complete an electronic diary
* Available for duration of study
* Negative pregnancy test for subjects in group 2 age 50 to 64 years
* Practice abstinence or use reliable birth control if age is 50 to 64 years

Exclusion Criteria:

* History of allergic reaction to any vaccine
* Previous vaccination with licensed or experimental pneumococcal vaccine
* S. pneumonia infection within past 5 years before investigational product administration
* Known or suspected immunodeficiency or received treatment including cytotoxic agents or systemic corticosteroids, serious chronic disorder such as malignancy cancer
* Receipt of plasma products or immunoglobulins within 60 days
* Bleeding conditions or diathesis
* Receipt of investigational product within 28 days before study entry
* Other severe acute or chronic medical or psychiatric condition

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2011-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- Mexico (4):
  - Instituto Mexicano de Investigación Clínica, S.A. de C.V, México, D.f.
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico City
  - Star Medica, Morelia, Michoacán
  - Hospital General de Durango, Durango

REFERENCES:
- [Derived] Tinoco JC, Juergens C, Ruiz Palacios GM, Vazquez-Narvaez J, Enkerlin-Pauwells HL, Sundaraiyer V, Pathirana S, Kalinina E, Gruber WC, Scott DA, Schmoele-Thoma B. Open-label trial of immunogenicity and safety of a 13-valent pneumococcal conjugate vaccine in adults >/= 50 years of age in Mexico. Clin Vaccine Immunol. 2015 Feb;22(2):185-92. doi: 10.1128/CVI.00711-14. Epub 2014 Dec 10. PMID 25499011
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1851048&StudyName=13-valent%20Pneumococcal%20Conjugate%20Vaccine%20Study%20in%20Adults%20%3D%3E%2050%20Years%20of%20Age%20in%20Mexico

RESULTS

PARTICIPANT FLOW:
Groups:
- 13vPnC, Cohort 1: Participants 50 to 64 years of age received 13-valent pneumococcal conjugate vaccine (13vPnC) administered as a 0.5 milliliter (mL) single dose intramuscularly on Day 1.
- 13vPnC, Cohort 2: Participants greater than or equal to (>=) 65 years of age received 13vPnC administered as a 0.5 mL single dose intramuscularly on Day 1.
Period: Overall Study
Arm/Group | 13vPnC, Cohort 1 | 13vPnC, Cohort 2
Started | 162 | 162
Vaccinated | 162 | 161
Completed | 160 | 161
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 13vPnC, Cohort 1 | 13vPnC, Cohort 2 | Total
Number analyzed (Participants) | 162 | 161 | 323
Age Continuous [Mean (Standard Deviation); unit: years] | 55.7 (4.0) | 73.4 (5.8) | 64.5 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 84 | 180
  Male | 66 | 77 | 143

OUTCOME MEASURES:

1. Primary Outcome: Serotype-Specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) 1 Month After Vaccination
Description: Serotype-specific OPA GMTs for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were determined in the blood samples of all the participants using a quantitative functional OPA assay. Confidence intervals (CIs) for GMT are back transformations of a CI based on the Student t distribution for the mean logarithm of the titers. Individual OPA assay values below the assay LLOQ (lower limit of quantification) were set at a titer of 0.5*limit of detection (LOD [8]) = (titer of 4) for the purpose of calculating the OPA GMT.
Time Frame: One month (28 to 42 days) after vaccination
Population: Evaluable Immunogenicity Population (EIP): eligible participants who received vaccine, had blood drawn within the pre-specified time frames, had at least 1 valid and determinate assay result for proposed analysis, received no prohibited vaccines, and had no other major protocol violations.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC, Cohort 1 | 13vPnC, Cohort 2
Number analyzed (Participants) | 155 | 159
titer
  1 | 120 [92.3 to 155.3] | 84 [62.8 to 112.5]
  3 | 88 [72.4 to 106.9] | 89 [70.8 to 111.5]
  4 | 1729 [1377.6 to 2170.9] | 1209 [977.1 to 1495.9]
  5 | 288 [208.6 to 398.3] | 285 [208.7 to 388.9]
  6A | 3380 [2732.9 to 4179.6] | 3343 [2625.2 to 4256.6]
  6B | 3982 [3273.2 to 4845.0] | 3384 [2708.6 to 4227.2]
  7F | 3130 [2660.9 to 3681.4] | 1929 [1564.7 to 2378.1]
  9V | 2416 [1901.0 to 3071.4] | 1402 [1030.8 to 1906.8]
  14 | 1569 [1267.9 to 1940.3] | 1316 [1068.9 to 1619.3]
  18C | 3063 [2405.9 to 3900.7] | 2197 [1727.2 to 2794.8]
  19A | 1542 [1257.9 to 1889.0] | 1196 [990.6 to 1443.1]
  19F | 1104 [828.1 to 1473.1] | 1188 [905.0 to 1558.6]
  23F | 879 [650.3 to 1187.7] | 930 [667.1 to 1296.2]

2. Primary Outcome: Percentage of Participants Reporting Pre-Specified Local Reactions Within 14 Days After Vaccination
Description: Local reactions reported using an electronic diary. Redness and Swelling scaled as Any (redness present or swelling present), Mild (2.5 to 5.0 centimeters [cm]), Moderate (5.1 to 10.0 cm), Severe (>10 cm). Pain at injection site scaled as Any (pain present), Mild (does not interfere with activity), Moderate (interferes with activity), Severe (prevents daily activity).
Time Frame: Within 14 days after vaccination
Population: Safety Population included all participants who received vaccine. N (Number of Participants Analyzed)=participants reporting yes for at least 1 day or no for all 14 days and n=participants reporting yes for at least 1 day or no for all 14 days for specified local reaction for each group respectively. Participants may be represented in >1 category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC, Cohort 1 | 13vPnC, Cohort 2
Number analyzed (Participants) | 152 | 139
percentage of participants
  Redness: Any (n=125, 120) | 14.4 [8.8 to 21.8] | 15.8 [9.8 to 23.6]
  Redness: Mild (n=124, 120) | 9.7 [5.1 to 16.3] | 13.3 [7.8 to 20.7]
  Redness: Moderate (n=125, 115) | 8.8 [4.5 to 15.2] | 7.0 [3.1 to 13.2]
  Redness: Severe (n=125, 112) | 2.4 [0.5 to 6.9] | 0.0 [0.0 to 3.2]
  Swelling: Any (n=130, 120) | 21.5 [14.8 to 29.6] | 13.3 [7.8 to 20.7]
  Swelling: Mild (n=127, 120) | 18.1 [11.8 to 25.9] | 11.7 [6.5 to 18.8]
  Swelling: Moderate (n=127, 114) | 8.7 [4.4 to 15.0] | 4.4 [1.4 to 9.9]
  Swelling: Severe (n=125, 113) | 2.4 [0.5 to 6.9] | 0.9 [0.0 to 4.8]
  Pain at injection site: Any (n=151, 137) | 75.5 [67.8 to 82.1] | 60.6 [51.9 to 68.8]
  Pain at injection site: Mild (n=151, 136) | 74.2 [66.4 to 80.9] | 60.3 [51.6 to 68.6]
  Pain at injection site: Moderate (n=130, 117) | 21.5 [14.8 to 29.6] | 8.5 [4.2 to 15.2]
  Pain at injection site: Severe (n=125, 113) | 3.2 [0.9 to 8.0] | 3.5 [1.0 to 8.8]

3. Primary Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events Within 14 Days After Vaccination
Description: Systemic events reported using electronic diary. Fever-Any:>=38 degrees Celsius (C), Mild (M):>=38 to <38.5 degrees C, Moderate(Mod):>=38.5 to <39 degrees C, Severe (S):>=39 to <=40 degrees C, Potentially life threatening:>40 degrees C. Headache, fatigue, muscle pain, joint pain- Any: present, M:did not interfere with activity, Mod:some interference, S:activity prevented. Vomiting- Any:present, M:1-2 times/day (d), Mod:>2/d, S:required intravenous hydration. Diarrhoea- Any:present, M:2-3 loose stools/d, Mod:4-5/d, S:>=6/d. All reports of fever >40 degrees C were confirmed as data entry errors.
Time Frame: Within 14 days after vaccination
Population: Safety Population included all participants who received vaccine. N (Number of Participants Analyzed)=participants reporting yes for at least 1 day or no for all 14 days and n=participants reporting yes for at least 1 day or no for all 14 days for specified systemic event for each group respectively. Participants may be represented in >1 category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC, Cohort 1 | 13vPnC, Cohort 2
Number analyzed (Participants) | 155 | 145
percentage of participants
  Fever: Any (n=126, 118) | 2.4 [0.5 to 6.8] | 10.2 [5.4 to 17.1]
  Fever: Mild (n=126, 113) | 1.6 [0.2 to 5.6] | 3.5 [1.0 to 8.8]
  Fever: Moderate (n=125, 113) | 0.8 [0.0 to 4.4] | 1.8 [0.2 to 6.2]
  Fever: Severe (n=124, 113) | 0.8 [0.0 to 4.4] | 1.8 [0.2 to 6.2]
  Fever: Potentially life threatening (n=124, 116) | 0.0 [0.0 to 2.9] | 4.3 [1.4 to 9.8]
  Fatigue: Any (n=144, 132) | 47.2 [38.9 to 55.7] | 38.6 [30.3 to 47.5]
  Fatigue: Mild (n=142, 130) | 39.4 [31.3 to 48.0] | 36.2 [27.9 to 45.0]
  Fatigue: Moderate (n=134, 125) | 26.9 [19.6 to 35.2] | 20.0 [13.4 to 28.1]
  Fatigue: Severe (n=126, 113) | 6.3 [2.8 to 12.1] | 5.3 [2.0 to 11.2]
  Headache: Any (n=140, 129) | 44.3 [35.9 to 52.9] | 32.6 [24.6 to 41.4]
  Headache: Mild (n=140, 128) | 39.3 [31.1 to 47.9] | 30.5 [22.6 to 39.2]
  Headache: Moderate (n=129, 119) | 18.6 [12.3 to 26.4] | 16.0 [9.9 to 23.8]
  Headache: Severe (n=126, 115) | 4.0 [1.3 to 9.0] | 5.2 [1.9 to 11.0]
  Vomiting: Any (n=125, 113) | 4.0 [1.3 to 9.1] | 1.8 [0.2 to 6.2]
  Vomiting: Mild (n=125, 113) | 3.2 [0.9 to 8.0] | 1.8 [0.2 to 6.2]
  Vomiting: Moderate (n=124, 113) | 1.6 [0.2 to 5.7] | 0.9 [0.0 to 4.8]
  Vomiting: Severe (n=124, 112) | 0.0 [0.0 to 2.9] | 0.0 [0.0 to 3.2]
  Diarrhea: Any (n=134, 120) | 26.1 [18.9 to 34.4] | 15.0 [9.1 to 22.7]
  Diarrhea: Mild (n=129, 120) | 23.3 [16.3 to 31.5] | 14.2 [8.5 to 21.7]
  Diarrhea: Moderate (n=129, 113) | 6.2 [2.7 to 11.9] | 1.8 [0.2 to 6.2]
  Diarrhea: Severe (n=125, 112) | 0.8 [0.0 to 4.4] | 0.9 [0.0 to 4.9]
  Muscle pain: Any (n=147, 132) | 60.5 [52.2 to 68.5] | 43.9 [35.3 to 52.8]
  Muscle pain: Mild (n=146, 129) | 59.6 [51.2 to 67.6] | 40.3 [31.8 to 49.3]
  Muscle pain: Moderate (n=132, 123) | 23.5 [16.5 to 31.6] | 19.5 [12.9 to 27.6]
  Muscle pain: Severe (n=125, 116) | 5.6 [2.3 to 11.2] | 6.0 [2.5 to 12.0]
  Joint pain: Any (n=139, 129) | 35.3 [27.3 to 43.8] | 33.3 [25.3 to 42.2]
  Joint pain: Mild (n=137, 127) | 30.7 [23.1 to 39.1] | 29.9 [22.1 to 38.7]
  Joint pain: Moderate (n=130, 123) | 13.1 [7.8 to 20.1] | 17.1 [10.9 to 24.9]
  Joint pain: Severe (n=125, 116) | 4.0 [1.3 to 9.1] | 5.2 [1.9 to 10.9]
  Use of medication to treat fever (n=129, 118) | 11.6 [6.7 to 18.5] | 13.6 [8.0 to 21.1]
  Use of medication to treat pain (n=130, 121) | 13.8 [8.4 to 21.0] | 12.4 [7.1 to 19.6]

4. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received vaccine without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial/prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between vaccination and up to 1 month (28 to 42 days) after vaccination that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Baseline up to 1 Month (28 to 42 days) after vaccination
Population: Safety Population included all participants who received the vaccine.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC, Cohort 1 | 13vPnC, Cohort 2
Number analyzed (Participants) | 162 | 161
percentage of participants
  AEs | 11.1 [6.7 to 17.0] | 6.2 [3.0 to 11.1]
  SAEs | 0.0 [0.0 to 2.3] | 1.2 [0.2 to 4.4]

5. Secondary Outcome: Percentage of Participants Achieving Serotype-Specific Opsonophagocytic Activity (OPA) Titer With at Least Lower Limit of Quantification (LLOQ) 1 Month After Vaccination
Description: Percentage of participants achieving OPA GMTs with at least LLOQ for 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F) determined in blood samples of all participants using microcolony OPA assay. Exact 2-sided CI based on observed proportion of participants. LLOQ for each serotype: 1=1:18, 3=1:12, 4=1:21, 5=1:29, 6A=1:37, 6B=1:43, 7F=1:210, 9V=1:345, 14=1:35, 18C=1:31, 19A=1:18, 19F=1:48, 23F=1:13.
Time Frame: One month (28 to 42 days) after vaccination
Population: EIP: eligible participants who received vaccine, had blood drawn within the pre-specified time frames, had at least 1 valid and determinate assay result for proposed analysis, received no prohibited vaccines, and had no other major protocol violations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC, Cohort 1 | 13vPnC, Cohort 2
Number analyzed (Participants) | 155 | 159
percentage of participants
  1 | 90.3 [84.5 to 94.5] | 81.0 [74.0 to 86.8]
  3 | 94.8 [90.0 to 97.7] | 90.1 [84.2 to 94.4]
  4 | 97.4 [93.4 to 99.3] | 98.7 [95.3 to 99.8]
  5 | 89.2 [83.0 to 93.7] | 90.8 [85.0 to 94.9]
  6A | 98.7 [95.4 to 99.8] | 98.1 [94.6 to 99.6]
  6B | 99.4 [96.4 to 100.0] | 98.7 [95.5 to 99.8]
  7F | 99.4 [96.5 to 100.0] | 97.5 [93.6 to 99.3]
  9V | 96.8 [92.6 to 98.9] | 92.3 [86.9 to 95.9]
  14 | 98.1 [94.4 to 99.6] | 98.1 [94.5 to 99.6]
  18C | 98.1 [94.4 to 99.6] | 98.7 [95.4 to 99.8]
  19A | 99.3 [96.4 to 100.0] | 99.4 [96.5 to 100.0]
  19F | 95.4 [90.7 to 98.1] | 96.0 [91.5 to 98.5]
  23F | 94.2 [89.2 to 97.3] | 91.7 [86.2 to 95.5]

6. Secondary Outcome: Serotype-Specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Fold Rise (GMFR) From Pre-Vaccination to 1 Month Post-Vaccination
Description: Geometric mean fold rises (GMFRs) for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) from pre-vaccination to 1 month post-vaccination were computed using the logarithmically transformed assay results. CIs for GMFR are back transformations of a CI based on the Student t distribution for the mean logarithm of the titers.
Time Frame: Pre-vaccination to 1 month (28 to 42 days) after vaccination
Population: EIP: eligible participants who received vaccine, had blood drawn within the pre-specified time frames, had at least 1 valid and determinate assay result, received no prohibited vaccines, and had no other major protocol violations. Here "N" signifies participants with valid and determinate assay results at both pre-vaccination and post-vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | 13vPnC, Cohort 1 | 13vPnC, Cohort 2
Number analyzed (Participants) | 153 | 158
fold rise
  1 | 21.3 [16.17 to 28.16] | 11.7 [8.70 to 15.82]
  3 | 12.5 [9.77 to 16.05] | 7.8 [6.03 to 10.02]
  4 | 57.7 [36.40 to 91.36] | 19.9 [13.23 to 29.88]
  5 | 37.3 [26.06 to 53.47] | 26.2 [18.74 to 36.72]
  6A | 62.3 [39.00 to 99.36] | 28.7 [19.76 to 41.70]
  6B | 18.1 [11.61 to 28.15] | 9.4 [6.61 to 13.45]
  7F | 43.2 [26.94 to 69.17] | 15.5 [10.05 to 23.80]
  9V | 8.8 [5.72 to 13.43] | 7.2 [4.72 to 10.98]
  14 | 5.3 [3.73 to 7.56] | 3.4 [2.58 to 4.56]
  18C | 44.3 [28.19 to 69.51] | 13.9 [9.21 to 21.09]
  19A | 30.0 [21.19 to 42.50] | 11.2 [7.99 to 15.69]
  19F | 42.8 [28.33 to 64.67] | 20.8 [13.38 to 32.29]
  23F | 63.6 [43.16 to 93.75] | 35.8 [24.16 to 52.95]

ADVERSE EVENTS:
Time Frame: Adverse events: recorded from signing of informed consent form to 28-42 days post 13vPnC. Participants recorded pre-specified AEs in electronic diary: local reactions and systemic events from Day 1 to 14 post 13vPnC.
Description: SAEs and AEs were grouped by system organ class and summarized. AEs included solicited AEs collected in the electronic diary (local and systemic reactions; systematic assessment) and unsolicited events collected on the case report form at each visit (nonsystematic assessment).
Arm/Group | 13vPnC, Cohort 1 | 13vPnC, Cohort 2
Serious Adverse Events (participants affected / at risk) | 0/162 | 2/161
Other Adverse Events (participants affected / at risk) | 119/162 | 88/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13vPnC, Cohort 1 (N=162) | 13vPnC, Cohort 2 (N=161)
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 13vPnC, Cohort 1 (N=162) | 13vPnC, Cohort 2 (N=161)
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 1 | 0
Influenza like illness (General disorders) | 0 | 1
Fever Any (General disorders) | 3/126 | 12/118
Fever Mild (General disorders) | 2/126 | 4/113
Fever Moderate (General disorders) | 1/125 | 2/113
Fever Severe (General disorders) | 1/124 | 2/113
Fever Potentially life threatening (General disorders) | 0/124 | 5/116 — All 'Fever Potentially life threatening' events were confirmed as data entry errors.
Fatigue Any (General disorders) | 68/144 | 51/132
Fatigue Mild (General disorders) | 56/142 | 47/130
Fatigue Moderate (General disorders) | 36/134 | 25/125
Fatigue Severe (General disorders) | 8/126 | 6/113
Headache Any (General disorders) | 62/140 | 42/129
Headache Mild (General disorders) | 55/140 | 39/129
Headache Moderate (General disorders) | 24/129 | 19/119
Headache Severe (General disorders) | 5/126 | 6/115
Vomiting Any (General disorders) | 5/125 | 2/113
Vomiting Mild (General disorders) | 4/125 | 2/113
Vomiting Moderate (General disorders) | 2/124 | 1/113
Vomiting Severe (General disorders) | 0/124 | 0/112
Diarrhea Any (General disorders) | 35/134 | 18/120
Diarrhea Mild (General disorders) | 30/129 | 17/120
Diarrhea Moderate (General disorders) | 8/129 | 2/113
Diarrhea Severe (General disorders) | 1/125 | 1/112
Muscle pain Any (General disorders) | 89/147 | 58/132
Muscle pain Mild (General disorders) | 87/146 | 52/129
Muscle pain Moderate (General disorders) | 31/132 | 24/123
Muscle pain Severe (General disorders) | 7/125 | 7/116
Joint pain Any (General disorders) | 49/139 | 43/129
Joint pain Mild (General disorders) | 42/137 | 38/127
Joint pain Moderate (General disorders) | 17/130 | 21/123
Joint pain Severe (General disorders) | 5/125 | 6/116
Gastroenteritis (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 0
Otitis media acute (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 2 | 0
Rhinitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Libido decreased (Psychiatric disorders) | 1 | 0
Urethral pain (Renal and urinary disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Redness Any (Skin and subcutaneous tissue disorders) | 18/125 | 19/120
Redness Mild (Skin and subcutaneous tissue disorders) | 12/124 | 16/120
Redness Moderate (Skin and subcutaneous tissue disorders) | 11/125 | 8/115
Redness Severe (Skin and subcutaneous tissue disorders) | 3/125 | 0/112
Swelling Any (Skin and subcutaneous tissue disorders) | 28/130 | 16/120
Swelling Mild (Skin and subcutaneous tissue disorders) | 23/127 | 14/120
Swelling Moderate (Skin and subcutaneous tissue disorders) | 11/127 | 5/114
Swelling Severe (Skin and subcutaneous tissue disorders) | 3/125 | 1/113
Pain at injection site Any (Skin and subcutaneous tissue disorders) | 114/151 | 83/137
Pain at injection site Mild (Skin and subcutaneous tissue disorders) | 112/151 | 82/136
Pain at injection site Moderate (Skin and subcutaneous tissue disorders) | 28/130 | 10/117
Pain at injection site Severe (Skin and subcutaneous tissue disorders) | 4/125 | 4/113
Hypertension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.